CLINICAL TRIAL: NCT00006981
Title: Phase I Study Of SS1(dsFv)-PE38 (SS1P) Anti-Mesothelin Immunotoxin in Advanced Malignancies: Continuous Infusion X 10 Days
Brief Title: Immunotoxin Therapy in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068351; NCI-01-C-0011; NCI-6249; NCT00006416 (obsolete NCT alias)
Record Dates: First submitted 2000-12-06; First posted 2003-01-27 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2005-05

CONDITIONS: Cervical Cancer; Fallopian Tube Cancer; Head and Neck Cancer; Lung Cancer; Malignant Mesothelioma; Ovarian Cancer; Pancreatic Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent non-small cell lung cancer; stage III cervical cancer; recurrent cervical cancer; stage IVB cervical cancer; stage IVA cervical cancer; squamous cell lung cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; advanced malignant mesothelioma; recurrent malignant mesothelioma; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent metastatic squamous neck cancer with occult primary; ovarian undifferentiated adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; cervical squamous cell carcinoma; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; fallopian tube cancer; primary peritoneal cavity cancer; ovarian carcinosarcoma; Brenner tumor; untreated metastatic squamous neck cancer with occult primary; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; ovarian mucinous cystadenocarcinoma; borderline ovarian surface epithelial-stromal tumor; ovarian sarcoma; ovarian stromal cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Fallopian Tube Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Mesothelioma, Malignant; Ovarian Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Squamous Cell Carcinoma of Head and Neck; Brenner Tumor; Salivary Gland Neoplasms | interventions — SS1(dsFv)PE38

INTERVENTIONS:
Biological: SS1(dsFv)-PE38 immunotoxin

SUMMARY:
RATIONALE: Immunotoxins can locate tumor cells and kill them without harming normal cells. Immunotoxin therapy may be an effective treatment for advanced cancer.

PURPOSE: Phase I trial to study the effectiveness of immunotoxins in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and toxic effects of SS1(dsFv)-PE38 immunotoxin in patients with advanced malignancies that express mesothelin.

Secondary

* Determine the response in patients treated with this drug.
* Determine the plasma pharmacokinetics of this drug in these patients.

OUTLINE: This is an open-label, dose-escalation study.

Patients receive SS1(dsFv)-PE38 immunotoxin IV continuously on days 1-10. Treatment repeats every 4 weeks for a maximum of 4 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of SS1(dsFv)-PE38 immunotoxin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy, including one of the following:

  * Malignant mesothelioma
  * Ovarian epithelial carcinoma (mucinous or nonmucinous), including primary peritoneal or fallopian tube carcinoma

    * Tumors that may have originated in the bowel (e.g., appendiceal carcinoma) and involve the ovary
    * Ovarian cancers of other histology are eligible provided they express mesothelin
  * Pancreatic cancer
  * Squamous cell lung cancer
  * Squamous cell cancer of the head and neck
  * Squamous cell cancer of the cervix
* Recurrent unresectable disease after prior standard anticancer therapy that was expected to prolong survival and improve quality of life OR unwilling to receive standard anticancer therapy
* At least 30% of initial or recurrent tumor cells positive (at least 1+) for mesothelin by immunohistochemistry
* Measurable or evaluable disease
* No known CNS or spinal cord involvement
* No clinically significant pericardial effusion

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN
* Albumin at least 3.0 g/dL
* Hepatitis B and C negative

Renal:

* Creatinine no greater than ULN OR
* Creatinine no greater than 2.0 mg/dL if creatinine clearance at least 50 mL/min
* Calcium no greater than ULN

Cardiovascular:

* No New York Heart Association class II-IV heart disease

Pulmonary:

* Oxygen saturation (SO_2) more than 92% on room air

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No detectable antibody to SS1(dsFv)-PE38
* No infection requiring parenteral antibiotics

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 week since prior hematopoietic growth factor therapy

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* At least 4 weeks since any prior antitumor therapy and recovered
* No other concurrent antitumor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kreitman, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Result] Kreitman RJ, Hassan R, Fitzgerald DJ, Pastan I. Phase I trial of continuous infusion anti-mesothelin recombinant immunotoxin SS1P. Clin Cancer Res. 2009 Aug 15;15(16):5274-9. doi: 10.1158/1078-0432.CCR-09-0062. Epub 2009 Aug 11. PMID 19671873
- [Result] Hassan R, Kreitman R, Strauss L, et al.: SS1(dsFv)-PE38 anti-mesothelin immunotoxin in advanced malignancies: phase I and pharmacokinetic study of alternate-day infusion. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-113, 2002.
- [Result] Kreitman R, Squires D, O'Hagan D, et al.: SS1(dsFv)-PE38 anti-mesothelin immunotoxin in advanced malignancies: phase I study of continuous infusion. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1896, 2002.